CLINICAL TRIAL: NCT03753893
Title: Prevalence of Ocular Manifestations in Inflammatory Rheumatic Diseases
Brief Title: Ocular Manifestations in Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Janet Pope, Professor of Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: MTJP001
Record Dates: First submitted 2018-10-31; First posted 2018-11-27 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Uveitis; Conjunctivitis; Keratoconjunctivitis Sicca; Xerophthalmia; Eye Hemorrhage; Optic Neuritis; Papilledema; Orbital Diseases; Retinal Vein Occlusion; Retinal Artery Occlusion; Macular Edema; Retinitis; Chorioretinitis; Iridocyclitis; Scleritis; Choroid Hemorrhage; Blindness; Amaurosis Fugax
MeSH Terms: conditions — Uveitis; Conjunctivitis; Keratoconjunctivitis Sicca; Xerophthalmia; Eye Hemorrhage; Optic Neuritis; Papilledema; Orbital Diseases; Retinal Vein Occlusion; Retinal Artery Occlusion; Macular Edema; Retinitis; Chorioretinitis; Iridocyclitis; Scleritis; Choroid Hemorrhage; Blindness; Amaurosis Fugax

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention used — no intervention used

SUMMARY:
This is a search strategy for determining the prevalence of ocular complications in inflammatory rheumatic diseases for the purposes of a meta analysis.

DETAILED DESCRIPTION:
For the purposes of determining the prevalence of ocular complications in inflammatory rheumatic diseases, the following search terms were used: conjunctivitis, keratoconjunctivitis sicca, xerophthalmia, uveitis, eye hemorrhage, optic neuritis, papilledema, orbital disease, retinal artery/vein occlusion, macular edema, retinitis, chorioretinitis, scleritis, iridocyclitis, choroid hemorrhage, blindness and amaurosis fugax.

These terms were searched in the context of a corresponding inflammatory disease on Medline, Cochrane and Web of Science from their inception (1966, 1991 and 1990 respectively) until the point of study completion.

Studies were included if they provided numerical data of the prevalence or incidence of ocular manifestations in an inflammatory rheumatic disease. Studies were excluded if they were review articles, case reports where all patients experienced the same ocular comorbidity, if different comorbidities were not grouped independently, and if the study reported on fewer than 20 patients. When the same study cohort was used in more than one analysis, the most recent or largest sample-size study was included. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) checklist was used to assess the quality of cohort, case-control, and cross-sectional studies.

ELIGIBILITY:
Inclusion Criteria:

* Studies were included if they provided numerical data of the prevalence or incidence of ocular manifestations in inflammatory rheumatic disease

Exclusion Criteria:

* review articles,
* case reports where all patients experienced the same ocular comorbidity
* if different comorbidities were not grouped independently
* if the study reported on fewer than 20 patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ocular involvement in inflammatory rheumatic disease
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of ocular manifestations of inflammatory rheumatic diseases | data is collected once per year up to 2020
  Prevalence of ocular manifestations of inflammatory rheumatic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Janet Pope, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No